CLINICAL TRIAL: NCT06140940
Title: Probing and Modulating Motor Imagery Capacities in Aphantasia
Brief Title: Motor Imagery in Aphantasia
Acronym: OLIPHANT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2023-A00887-38
Record Dates: First submitted 2023-11-13; First posted 2023-11-21 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Aphasia
MeSH Terms: conditions — Aphasia

STUDY DESIGN:
Intervention Model Description: Single-center prospective randomized, double-blind, sham-controlled, crossover study with two conditions: active tDCS + mental training and sham tDCS + mental training. A control group (participants with typical mental imagery abilities) will also be included for comparison at baseline.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants and experimenters (including tDCS operator) will not be informed about the nature (active or placebo) of the stimulation they will receive
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active stimulation group: 20 participants with aphantasia will receive a session of active HD-tDCS (Experimental): Participants will receive a session of active HD-tDCS at a current intensity of 4 mA for a duration of 15min. The placement of electrodes will be determined to specifically target the primary motor cortex (4 x 1 montage with the anode over C4). During the stimulation, participants will be engaged in a mental training task (sequential finger tapping-task).
  Interventions: Procedure: High-definition transcranial direct current (HD-tDCS), active condition
- placebo stimulation group: 20 participants with aphantasia will receive a session of sham HD-tDCS (Placebo Comparator): High-definition transcranial direct current (HD-tDCS), sham condition. Participants will receive a session of sham HD-tDCS, which will be delivered following the same procedures as active HD-tDCS but the intensity of the current will be set at 4mA during the 30 first seconds at the beginning of the 15-min period of the stimulation, and equal to 0 mA for the reminding period of stimulation to simulate the tingling sensation often experienced by individuals during active stimulation.
  The placement of electrodes will be determined to specifically target the primary motor cortex (4 x 1 montage with the anode over C4). During the stimulation, participants will be engaged in a mental training task (sequential finger tapping-task).
  Interventions: Procedure: High-definition transcranial direct current (HD-tDCS), sham condition

INTERVENTIONS:
Procedure: High-definition transcranial direct current (HD-tDCS), active condition — Participants will receive a session of active HD-tDCS at a current intensity of 4 mA for a duration of 15min. The placement of electrodes will be determined to specifically target the primary motor cortex (4 x 1 montage with the anode over C4). During the stimulation, participants will be engaged in a mental training task (sequential finger tapping-task).
  Arms: active stimulation group: 20 participants with aphantasia will receive a session of active HD-tDCS
Procedure: High-definition transcranial direct current (HD-tDCS), sham condition — Participants will receive a session of sham HD-tDCS, which will be delivered following the same procedures as active HD-tDCS but the intensity of the current will be set at 4mA during the 30 first seconds at the beginning of the 15-min period of the stimulation, and equal to 0 mA for the reminding period of stimulation to simulate the tingling sensation often experienced by individuals during active stimulation.
  The placement of electrodes will be determined to specifically target the primary motor cortex (4 x 1 montage with the anode over C4). During the stimulation, participants will be engaged in a mental training task (sequential finger tapping-task).
  Arms: placebo stimulation group: 20 participants with aphantasia will receive a session of sham HD-tDCS

SUMMARY:
The present study aims to characterize and modulate motor imagery abilities in individuals with aphantasia. The investigators will characterize the neurophysiological and physiological underpinnings of mental imagery abilities in participants with aphantasia by investigating several indices of motor imagery abilities and comparing them to participants with typical mental imagery abilities. The investigators will investigate whether non-invasive brain stimulation applied to the primary motor cortex improves mental imagery abilities in participants with aphantasia.

DETAILED DESCRIPTION:
The investigators will recruit 20 participants with aphantasia and 20 participants with typical mental imagery capacities (no-aphantasia groups). Participants in both groups will complete a 3-hour visit for inclusion and baseline measurements (Visit 1) which will include neurophysiological, autonomic nervous system, cognitive and behavioral measures.

Participants in the aphantasia group will complete 2 additional visits to receive active and sham tDCS sessions (Visit 2 and 3), according to a randomized, double-blind, sham-controlled, crossover design. Mental training will be done concurrently with tDCS using a sequential finger tapping-task (Truong et al., 2022). Participants will receive the instructions of trying to imagine themselves performing the motor task, by feeling their fingers moving as if they were actually moving it (kinesthetic modality of motor imagery).

Visits will be separated by at least 7 days.

ELIGIBILITY:
Inclusion Criteria:

* For the aphantasia group only: congenital aphantasia defined as a life-long inability to generate mental imagery (confirmed by a total score of 32 or less on the VVIQ, which is the gold standard questionnaire for aphantasia)
* For the no-aphantasia group only: typical mental imagery capacities (confirmed by a total score of more than 32 on the VVIQ)
* Covered by public health insurance
* Understanding the French language
* Signed written informed consent after being informed about the study

Exclusion Criteria:

* Presence or history of a somatic, neurologic, or mental illness
* Actual pain or musculoskeletal disorders at the upper limb
* Having a regular musical activity (more than once a week) because of high manual dexterity
* Contraindication for noninvasive brain stimulation including the presence of ferromagnetic or magnetic sensitive metal objects implanted in the head or in close proximity (e.g., brain stent, clip, cochlear implants, or stimulator)
* Pregnancy (controlled by urine pregnancy test in females without reported contraception)
* Active seizure disorder or history of seizures
* Participants under curatorship/guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-28 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Gains in motor performance following mental training | 2 times: immediately before tDCS (baseline) and immediately after tDCS
  Gains in motor performance following mental training combined with tDCS will be measured using a sequential finger tapping-task. Gains following training will be expressed as a percentage of the baseline performance.

SECONDARY OUTCOMES:
Motor corticospinal excitability at rest and during kinesthetic motor imagery | 1 time at baseline (Visit 1), in both groups
  Motor corticospinal excitability will be assessed with single-pulse transcranial magnetic stimulation (TMS) applied over the primary motor cortex representation of the non-dominant hand. Using electromyography, we will measure the peak-to-peak mean amplitude of motor evoked potentials (MEPs, measured in mV) in the contralateral first dorsal interosseous muscle both at rest and during kinesthetic motor imagery.
Heart rate variability | through study completion, an average of 1 month
  Heart rate variability, including respiratory sinus arrhythmia measures, expressed in milliseconds (ms), will be assessed at rest and during kinesthetic motor imagery by recording the heart rate using three electrodes placed in the left chest area. These electrodes will be connected to the Biopac MP150 system and monitored with the Acqknowledge software
Skin conductance | through study completion, an average of 1 month
  Amplitude of electrodermal response will be measured at rest, during actual movements and during kinesthetic motor imagery using the Biopac MP150 system with the Acqknowledge software. The ratio between amplitudes during imagined/actual movements will be computed (expressed in percent).
Mental imagery abilities | 1 time at baseline, in both groups
  Mental imagery abilities in different sensory modalities will be measured as scores at the following questionnaires: Vividness of Visual Imagery Questionnaire (VVIQ; range 16-80)
Mental imagery abilities | 1 time at baseline, in both groups
  Mental imagery abilities in different sensory modalities will be measured as scores at the following questionnaires: the Kinesthetic and Visual Imagery Questionnaire (KVIQ; range 20-100).
Mental imagery abilities | 1 time at baseline, in both groups
  Mental imagery abilities in different sensory modalities will be measured as scores at the following questionnaires: the Movement Imagery Questionnaire-Revised (MIQ-R; range 14-98)
Mental imagery abilities | 1 time at baseline, in both groups
  Mental imagery abilities in different sensory modalities will be measured as scores at the following questionnaires: the Test of Ability in Movement Imagery (TAMI; range 0-24)
Mental imagery abilities | 1 time at baseline, in both groups
  Mental imagery abilities in different sensory modalities will be measured as scores at the following questionnaires: Plymouth Sensory Imagery Questionnaire (Psi-Q; range 0-70)
Source monitoring performance | 1 time at baseline, in both groups
  Source monitoring performance will be evaluated using a specific source monitoring task . Source-monitoring accuracy scores (range 0-100) will be calculated as proportions of accurate source attributions for each source
Implicit motor imagery capacities | 1 time at baseline, in both groups
  Implicit motor imagery capacities will be measured using a hand laterality judgment task . The percentage of correct response at the task will be calculated (range 0-100%).
Performance of time-to-contact estimation | 1 time at baseline, in both groups
  Performance will be measured using a specific time-to-contact (TTC) task. A TTC task involves temporal prediction in that the task requires a participant to predict the moment at which an event will occur given past sensory information (e.g., an auditory stimuli). The estimation of TTC requires determining the moment of contact (TTCa). The analysis of performance is based on BIAS quantification, which measures the average difference between individual estimation and TTCa

CONTACTS AND LOCATIONS:
Overall Officials: Marine MONDINO, PhD, Principal Investigator — CH le Vinatier
Locations (1):
- Centre Hospitalier le Vinatier, Bron, France

IPD SHARING:
Plan to Share IPD: No